CLINICAL TRIAL: NCT06834152
Title: Online Adaptive Stereotactic Body Radiotherapy for Localized Prostate Cancer in Patients With Lower Urinary Tract Symptoms and/or Prostate Hyperplasia (X-SMILE)
Brief Title: Online Adaptive Stereotactic Body Radiotherapy for Localized Prostate Cancer (X-SMILE)
Acronym: X-SMILE
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: RAO-24-014
Record Dates: First submitted 2025-02-06; First posted 2025-02-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Localized Prostate Carcinoma; Prostate Cancer (Adenocarcinoma); Prostate Hyperplasia; Lower Urinary Track Symptoms
Keywords: radiotherapy; SBRT; MRI; CT; stereotactic radiotherapy; localized prostate cancer; lower urinary tract symptoms; prostate hyperplasia; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pilot study: For our pilot study, we assumed that around 3% of patients would have grade 3 acute urogenital toxicity (i.e. 1 patient). The rate of treatment discontinuation within 3 months was considered negligible. Our aim was to show with high probability, that the event rate was below a clinically acceptable threshold, which was set at 20%. Under the null hypothesis, this design with an alpha of 0.05 and power of 80% results in an expected number of cases of 30. Dropouts prior to treatment start will be replaced.
  Interventions: Radiation: radiotherapy
- Validation Cohort: For our validation study, we assume that around 3% of patients will have grade 3 long-term urogenital toxicity (i.e. 2 patients). The rate of treatment discontinuation within 3 months is considered negligible. Our aim is to show with high probability, that the event rate is below a clinically acceptable threshold, which is set at 12%. Under the null hypothesis, this design with an alpha of 0.05 and power of 80% results in an expected number of cases of 75. Dropouts prior to treatment start will be replaced.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Patients with prostate cancer in the medium or high risk range who are planned to receive definitive CT or MRI-adaptive SBRT.

SUMMARY:
The aim of this phase II international multicenter study is to evaluate the safety, feasibility, and efficacy of CT or MRI-adaptive SBRT, delivered in five weekly fractions, in patients with newly diagnosed localized prostate cancer who have lower urinary tract symptoms and/or prostatic hyperplasia.

DETAILED DESCRIPTION:
Background: Stereotactic body radiotherapy (SBRT) for localized prostate cancer has demonstrated non-inferior oncological outcomes and toxicity profiles to conventionally or moderately hypofractioned radiotherapy regimens, while offering the advantage of shorter treatment durations. However, SBRT may not be suitable for all patients, particularly those with lower urogenital tract symptoms and/or prostatic hyperplasia.

Methods: This study aims to evaluate the safety and efficacy of weekly computed tomography (CT) or magnetic resonance image-guided (MRI) online adaptive SBRT in patients with intermediate to (very) high-risk localized prostate cancer who present with lower urinary tract symptoms (International Prostate Symptom Score [IPSS] > 12) and/or have prostate hyperplasia (prostate volume >60 mL). The primary outcome measure is urogenital toxicity grade ≥3 within 3 months after completion of SBRT (according to CTCAE V5.0 and RTOG) or discontinuation of therapy. Our aim is to show that the event rate is at 3% below a clinically acceptable threshold, which is set at 20%. Under the null hypothesis, this design with an alpha of 0.05 and power of 80% results in an expected number of cases of 30. In our validation cohort we assume that around 3% of patients will have grade 3 long-term urogenital toxicity (i.e. 2 patients). The rate of treatment discontinuation within 3 months is considered negligible. Our aim is to show with high probability, that the event rate is below a clinically acceptable threshold, which is set at 12%. Under the null hypothesis, this design with an alpha of 0.05 and power of 80% results in an expected number of cases of 75.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed localized prostate cancer
* planned treatment is SBRT according to standard of care and consists of definitive CT or MRI online adaptive SBRT of the prostate according to the PACE trial which includes a total dose to clinical target volume 1 (CTV1, i.e. prostate and proximal 1 cm of the seminal vesicle) of 40.0 Gy in 5 weekly fractions (single dose of 8.0 Gy) and total dose to planning target volume 1 (PTV1) of 37.5 Gy in 5 weekly fractions (single dose of 7.5 Gy) with a compromise for bowel sparing allowed. For patients with unfavorable intermediate to very high-risk disease (according to NCCN guidelines) a total dose to the planning target volume 2 (PTV2, i.e. proximal 1-2 cm of the seminal vesicle) of 32.5 Gy in 5 weekly fractions (single dose of 6.5 Gy) will be delivered.
* intermediate to (very) high risk localized prostate cancer (≤ cT3a and Gleason score ≤ 9 and/or PSA ≤ 20 ng/ml)
* prostate volume > 60 cc and/or IPSS > 12;

Exclusion Criteria:

* Very high risk localized prostate cancer with indication for ADT and ARPI (i.e. Gleason ≥ 8 and cT3a)
* Involvement of seminal vesicles (cT3b)
* Contraindications against definitive CT or MRI-adaptive radiotherapy of the prostate, e.g. inflammatory bowel disease (IBD); previous radiotherapy in the pelvis, previous local radiotherapy of the prostate, contraindication for MRI or CT;
* Patients with severe genitourinary symptoms (e.g. recent urinary retention ≥ grade 3 according CTCAE v.5.0);
* Lymph node metastases or distant metastases (i.e. no localised prostate cancer);
* Participation in a clinical trial which might influence the results of this project.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This international multicenter prospective phase II study, conducted in collaboration with several academic hospitals in Switzerland and Germany, will include patients with histologically confirmed intermediate to (very) high risk localized prostate cancer with lower urinary tract symptoms and/or prostate hyperplasia. These patients are planned to receive weekly CT or MRI online adaptive SBRT for localized prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
acute grade ≥ III urogenital toxicity | ≤ 3 months after completion of radiotherapy
  The primary endpoint is acute grade ≥ III urogenital toxicity ≤3 months after completion of radiotherapy (according to the NCI CTCAE V5 or RTOG) or treatment discontinuation related to treatment.

SECONDARY OUTCOMES:
Gastrointestinal toxicity of grade ≥3 | ≤ 3 months after completion of radiotherapy
  Gastrointestinal toxicity of grade ≥3 within 3 months after completion of radiotherapy (according to CTCAE V5.0 and RTOG)
Mortality | ≤1 year after initiation of radiotherapy
  Mortality (related to treatment and/or disease).
Urogenital and gastrointestinal toxicities | ≤ 5 years after completion of radiotherapy
  Number of urogenital and gastrointestinal toxicities within 5 years after completion of radiotherapy and their severity.
Biochemical progression-free survival | ≤ 5 years after completion of radiotherapy
  Biochemical progression-free survival (determined from the start of therapy until the occurrence of PSA recurrence according to the Phoenix criteria i.e. post- therapeutic PSA nadir + 2 ng/ml),
Hormonal therapy-free survival | ≤ 5 years after completion of radiotherapy
  Hormonal therapy-free survival (determined from the start of therapy until the start of hormonal therapy,
Overall survival | 5 years after completion of radiotherapy
  overall survival (defined from the start of therapy until death or censoring)
Quality-of-life questionnaire C-30 from the European Organisation for Research and Treatment of Cancer | ≤ 5 years after completion of radiotherapy
  Quality-of-life measured using the EORTC QLQ-C30 questionnaire during and after treatment
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Uroflowmetry (optional) | Uroflowmetry ≤ 6 weeks prior to the start of radiotherapy
  Uroflowmetry prior to the start of radiotherapy (optional study procedure)
Quality-of-life questionnaire PR25 of the European Organisation for Research and Treatment of Cancer | ≤ 5 years after completion of radiotherapy
  Quality-of-life measured using the QLQ-PR25 questionnaire during and after treatment
  All of the scales and single-item measures range in score from 0 to 100. A high score for the Sexual Activity and Sexual Functioning scales represents a high level of functioning, whereas a high score for the Urinary, Bowel, and Hormonal Treatment-Related symptoms scales and Incontinence Aid item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Prof. Dr. med., Study Chair — University of Zurich; Tiuri E. Kroese, MD, PhD, Principal Investigator — University of Zurich; Matthias Guckenberger, Principal Investigator — University of Zurich
Locations (3):
- Germany (2):
  - Klinik für Radioonkologie und Strahlentherapie, Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinik und Poliklinik für Strahlentherapie und Radioonkologie, Universitätsklinikum LMU, Munich, Bavaria
- University Hospital Zurich, Department of Radio-Oncology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this trial after de-identification. Other documents may be shared include the study protocol.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months after article publication.
Access Criteria: Proposals to access study data should send request to matthias.guckenberger@usz.ch. To gain access, data requesters must sign data access agreement.

REFERENCES:
- [Derived] Kroese T, Andratschke N, Belka C, Corradini S, Marschner S, Liermann J, Horner-Rieber J, Fink C, Debus J, Silvia F, Tanadini-Lang S, Pouymayou B, Mencarelli A, Fesslmeier D, Schiess A, Guckenberger M, Mayinger M. Online adaptive stereotactic body radiotherapy for localized prostate cancer in patients with lower urinary tract symptoms and/or prostate hyperplasia (X-SMILE). Radiat Oncol. 2025 May 28;20(1):90. doi: 10.1186/s13014-025-02653-4. PMID 40437508